CLINICAL TRIAL: NCT03700593
Title: Feasibility and Safety of Single Port Robot in Colorectal Procedures
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Marks Colorectal Surgical Associates (Other)
Responsible Party: Principal Investigator, Dr. John Marks, Chief of Colorectal Surgery, Marks Colorectal Surgical Associates
Other Study IDs: F/N-R19-3864L
Record Dates: First submitted 2018-10-02; First posted 2018-10-09 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Colon Cancer; Colon Polyp; Rectal Cancer; Diverticulitis; Prolapse, Rectal; Rectal Polyp; Inflammatory Bowel Diseases
Keywords: Single port robotic surgery; Minimally invasive colectomy; Single port robotic colectomy; Single port robotic TEM
MeSH Terms: conditions — Colonic Neoplasms; Colonic Polyps; Rectal Neoplasms; Diverticulitis; Rectal Prolapse; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Single Port Robotic Colorectal Surgery Patients: All patients who undergo a single port robot colorectal surgery.
  Interventions: Device: Single Port Robotic Colorectal Surgery

INTERVENTIONS:
Device: Single Port Robotic Colorectal Surgery — Single Port Robotic Colorectal Surgery

SUMMARY:
The purpose of this study is to evaluate the safety and feasibility of using the Single Port (SP) robot (daVinci, Intuitive Surgical) to perform single port robotic colon surgery and transanal robotic surgery. The hypothesis of the study is that the SP robot will prove a safe effective modality to perform these procedures.

DETAILED DESCRIPTION:
In the colorectal arena, the robotic approach for benign and malignant disease is well established, with a great deal of literature generated regarding the safety and benefits of a colorectal robotic approach for benign and malignant disease. The section of colorectal surgery at the Lankenau Medical Center has been an active and robust contributor to surgical literature on laparoscopic surgery, robotic colorectal surgery, and single port laparoscopic surgery. Its one investigator has been involved in the development of clinical applications to the single port robotic platform where this has been utilized in cadaver work that has been published. Recently, the SP robot has gone through FDA clearance and is now available for clinical utilization. The FDA approval is for urologic surgery. The SP robot will be utilized in the same fashion to perform the same colorectal operations that the investigators have been performing with multiple port placements in the past to accomplish robotic surgery in a single port platform in the colorectal arena. The principal investigator has worked on the SP robot over the past 3 years with extensive cadaver experience to develop its safe application in the colorectal field. This study will entail a collection of demographics, preoperative, perioperative and postoperative outcomes of the patients into a database to follow this, report on the outcomes, and notably answer questions to demonstrate the feasibility and safety of this approach in colorectal patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients being considered for minimally invasive colorectal surgery will be evaluated for participation in the study.

Exclusion Criteria:

* emergency surgery
* inability to offer informed consent
* pregnant patients

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients with a colorectal pathology requiring a minimally invasive colorectal procedure.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-10-15 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the SP robot | 30 days
  Calculating the percentage of cases successfully performed using the SP robot, without conversion.
Rate of postoperative complications and mortality of the SP robot | 30 days
  Measuring the post-operative morbidity and mortality will be used to evaluate the safety of the SP robot.

SECONDARY OUTCOMES:
Assessment of patients quality of life using validated questionnaires. | 1 year
  Validated questionnaire will be administered to assess the quality of life of patients:
  - RAND 36 item Health Survey (by the RAND corporation): All items are scored so that a high score defines a more favorable health state. In addition, each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively. This validated questionnaire asks patients to rate their own health and rate their ability to perform a variety of everyday activities using the same scale.
Assessment of patients' satisfaction with their surgical scars using validated questionnaires. | 1 year
  Validated questionnaire will be administered to assess the patients satisfaction with surgery Patient Scar Assessment Questionnaire (PSAQ)- The PSAQ consists of 5 subscales: Appearance (# of items-9; min-9; max-36), Consciousness (#-6; min-6; max-24), Satisfaction with Appearance (#-8; min-8; max-32) and Satisfaction with Symptoms (#-5; min-5; max-20). Higher scores define more favorable scar appearance, less consciousness of one's scar, increased satisfaction with appearance and symptoms. The scales for each of these subsections is the same; however, min and max scores differ due to differing numbers of questions in each section.
Assessment of patient's quality of recovery | 1 year
  - Quality of Recovery 40 questionnaire: score range: 40-200. Higher values represent better outcomes. The validate questionnaire measure quality of recovery by evaluating patients' comfort, emotions, physical independence, and support using the same scale.
Assessment of patients' postoperative body image satisfaction | 1 year
  Body image questionnaire- 13 items total; min score-13 and max score-100. Higher scores correlate to more favorable body image. In reflecting on their own body image, patients are then asked to rate how likely they would be to undergo a laparoscopic, open, versus single port surgery given their experience. These variables are measured on the same scale.

CONTACTS AND LOCATIONS:
Overall Officials: John H Marks, MD, Principal Investigator — Main Line Health System / Lankenau Medical Center
Locations (1):
- Lankenau Medical Center, Marks Colorectal Surgical Associates, Wynnewood, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marks JH, Agarwal S, Kunkel E, Schoonyoung H, Salem JF. Video Demonstration of an Initial Single-Port Robotic Transanal Total Mesorectal Excision. Dis Colon Rectum. 2021 Aug 1;64(8):e472-e473. doi: 10.1097/DCR.0000000000002139. No abstract available. PMID 34001710
- [Derived] Marks JH, Kunkel E, Salem JF, Martin CT, Anderson B, Agarwal S. First Clinical Experience With Single-Port Robotic Transanal Minimally Invasive Surgery: Phase II Trial of the Initial 26 Cases. Dis Colon Rectum. 2021 Aug 1;64(8):1003-1013. doi: 10.1097/DCR.0000000000001999. PMID 34001709

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2018-09-24): https://cdn.clinicaltrials.gov/large-docs/93/NCT03700593/Prot_ICF_000.pdf